CLINICAL TRIAL: NCT02357589
Title: 3 Versus 2 Dimensional HD Laparoscopy in Cholecystectomy: a Prospective, Single Blinded, Randomized, Controlled Trial
Brief Title: 3D vs 2D HD Laparoscopy in Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Hanna Koppatz, MD, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUCH-328-150127
Record Dates: First submitted 2015-02-03; First posted 2015-02-06 (Estimated); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Cholecystolithiasis
Keywords: 3D; laparoscopy; cholecystectomy
MeSH Terms: conditions — Cholecystolithiasis

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- 2D laparoscopic cholecystectomy (Active Comparator): The normal laparoscopic cholecystectomy with two dimensional view
  Interventions: Procedure: 2D laparoscopic cholecystectomy
- 3D laparoscopic cholecystectomy (Experimental): The normal laparoscopic cholecystectomy with three dimensional view
  Interventions: Procedure: 3D laparoscopic cholecystectomy

INTERVENTIONS:
Procedure: 2D laparoscopic cholecystectomy
  Arms: 2D laparoscopic cholecystectomy
Procedure: 3D laparoscopic cholecystectomy
  Arms: 3D laparoscopic cholecystectomy

SUMMARY:
The 3D-systems have emerged also to the world of surgery, and the three-dimensional laparoscopic systems are gradually entering the operating rooms. In the normal laparoscopy there are only two-dimensional view, which is somewhat challenging when operating in three-dimensional environment. Even though the 3D-systems have been widely studied in laboratory circumstances, there are still no evidence of benefits of 3D vs 2D in clinical point of view and no prospective randomized trials have been published. Therefore, the purpose of this study is to investigate is there something to gain in changing into 3D laparoscopic system for cholecystectomy (LCC).

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for laparoscopic cholecystectomy

Exclusion Criteria:

* Some other surgical operation planned during LCC
* Expected major risk of conversion (e.g. multiple previous abdominal operation, previous peritonitis, previous cholecystitis)
* Operating surgeon experience less than 5 3D laparoscopy operations

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2015-01; Primary Completion 2017-05-10 (Actual); Study Completion 2017-05-10 (Actual)

PRIMARY OUTCOMES:
Duration of surgery | Expected average time of surgery 1 hour

SECONDARY OUTCOMES:
Need for conversion into open surgery | During the operation, expected average time of surgery 1 hour
Intraoperative complications | During the operation, expected average time of surgery 1 hour
  Any complication during the operation e.g. hemorrhagic, liver, intestine or gallbladder rupture
Complications, Clavien-Dindo classification | 30 days after randomization
Postoperative stay in hospital | Expected range 0-7 day
Bleeding | During the operation, expected average time of surgery 1 hour
Number of participants with readmission(s) | 30 days after randomization
Total need of opioids in milligrams | Expected range 0-7 day
Mortality | 30 days after randomization
Operation theatre time | Expected average 1,5 hours
Postoperative pain, VAS | Expected range 0-7 day

OTHER OUTCOMES:
Incisional hernias | after 1, 5 and 10 year

CONTACTS AND LOCATIONS:
Overall Officials: Ville Sallinen, MD, PhD, Study Chair — Helsinki University Central Hospital
Locations (1):
- Helsinki University Central Hospital, Helsinki, Finland

REFERENCES:
- [Derived] Koppatz H, Harju J, Siren J, Mentula P, Scheinin T, Sallinen V. Three-dimensional versus two-dimensional high-definition laparoscopy in cholecystectomy: a prospective randomized controlled study. Surg Endosc. 2019 Nov;33(11):3725-3731. doi: 10.1007/s00464-019-06666-5. Epub 2019 Feb 1. PMID 30710315